CLINICAL TRIAL: NCT05544786
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, CROSSOVER STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF NIRMATRELVIR (PF-07321332) /RITONAVIR ORAL POWDER IN 3 DIFFERENT FOOD DELIVERY VEHICLES RELATIVE TO THE NIRMATRELVIR (PF-07321332) /RITONAVIR COMMERCIAL TABLETS UNDER FASTED CONDITIONS, AND THE EFFECT OF FOOD ON RELATIVE BIOAVAILABILITY OF NIRMATRELVIR (PF-07321332) /RITONAVIR ORAL POWDER IN HEALTHY ADULT PARTICIPANTS
Brief Title: Relative Bioavailability Study of Nirmatrelvir/Ritonavir Oral Powder Relative to the Commercial Tablets and Estimation of the Effect of Food on Bioavailability of the Nirmatrelvir/Ritonavir Oral Powder in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671036; 2022-002497-86 (EudraCT Number)
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-11

CONDITIONS: Biological Availability
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Nirmatrelvir; Paxlovid
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: Nirmatrelvir/ritonavir (Active Comparator): Nirmatrelvir and ritonavir tablets
  Interventions: Drug: Nirmatrelvir/ ritonavir
- Treatment B: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ritonavir with water
  Interventions: Drug: Nirmatrelvir/Ritonavir
- Treatment C: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir with infant formula
  Interventions: Drug: Nirmatrelvir/Ritonavir
- Treatment D: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir with vanilla pudding
  Interventions: Drug: Nirmatrelvir/ritonavir
- Treatment E: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir with food and vanilla pudding
  Interventions: Drug: Nirmatrelvir/ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir/ ritonavir — Single oral dose of nirmatrelvir/ritonavir tablets under fasted condition
  Arms: Treatment A: Nirmatrelvir/ritonavir
Drug: Nirmatrelvir/Ritonavir — Single oral dose of nirmatrelvir/ritonavir mixed in water under fasted condition
  Arms: Treatment B: Nirmatrelvir/ ritonavir
Drug: Nirmatrelvir/Ritonavir — Single oral dose of nirmatrelvir/ritonavir mixed in infant formula under fasted condition
  Arms: Treatment C: Nirmatrelvir/ ritonavir
Drug: Nirmatrelvir/ritonavir — Single oral dose of nirmatrelvir/ritonavir mixed in vanilla pudding under fasted condition
  Arms: Treatment D: Nirmatrelvir/ ritonavir
Drug: Nirmatrelvir/ritonavir — Single oral dose of nirmatrelvir/ritonavir mixed in vanilla pudding under fed condition
  Arms: Treatment E: Nirmatrelvir/ ritonavir

SUMMARY:
The purpose of this study is to estimate the relative bioavailability (rBA) of nirmatrelvir/ritonavir oral powder in 3 different food vehicles relative to the Paxlovid® tablets under fasted condition in healthy adult participants, and to estimate the effect of food on the rBA of the nirmatrelvir/ritonavir oral powder formulation. The study will also assess the safety, tolerability, and palatability of nirmatrelvir/ritonavir oral powder in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination (PE), laboratory tests, vital signs and standard 12 lead ECGs.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than New York Heart Association (NYHA) 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antibody (HCVAb). Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Participant who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants were assigned to the study.
Groups:
- Treatment A->B->C->D->E: Each enrolled participant participated in 5 study periods (1-5) to receive 5 different treatments (A, B, C, D, E) according to the sequence determined by randomization. Between each treatment, a minimum of 4 days washout was proposed to minimize any residual nirmatrelvir concentrations prior to start of the next treatment.
  Period 1: Treatment A: Single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted condition.
  Period 2: Treatment B: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in water under fasted condition.
  Period 3: Treatment C: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in infant formula under fasted condition.
  Period 4: Treatment D: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition.
  Period 5: Treatment E: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition.
- Treatment B->C->A->D->E: Each enrolled participant participated in 5 study periods (1-5) to receive 5 different treatments (A, B, C, D, E) according to the sequence determined by randomization. Between each treatment, a minimum of 4 days washout was proposed to minimize any residual nirmatrelvir concentrations prior to start of the next treatment.
  Period 1: Treatment B: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in water under fasted condition.
  Period 2: Treatment C: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in infant formula under fasted condition.
  Period 3: Treatment A: Single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted condition.
  Period 4: Treatment D: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition.
  Period 5: Treatment E: Single oral dose of nirmatrelvir 300 and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition.
- Treatment C->A->B->D->E: Each enrolled participant participated in 5 study periods (1-5) to receive 5 different treatments (A, B, C, D, E) according to the sequence determined by randomization. Between each treatment, a minimum of 4 days washout was proposed to minimize any residual nirmatrelvir concentrations prior to start of the next treatment.
  Period 1: Treatment C: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in infant formula under fasted condition.
  Period 2: Treatment A: Single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted condition.
  Period 3: Treatment B: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in water under fasted condition.
  Period 4: Treatment D: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition.
  Period 5: Treatment E: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition.
- Treatment A->C->B->E->D: Each enrolled participant participated in 5 study periods (1-5) to receive 5 different treatments (A, B, C, D, E) according to the sequence determined by randomization. Between each treatment, a minimum of 4 days washout was proposed to minimize any residual nirmatrelvir concentrations prior to start of the next treatment.
  Period 1: Treatment A: Single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted condition.
  Period 2: Treatment C: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in infant formula under fasted condition.
  Period 3: Treatment B: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in water under fasted condition.
  Period 4: Treatment E: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition.
  Period 5: Treatment D: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition.
- Treatment B->A->C->E->D: Each enrolled participant participated in 5 study periods (1-5) to receive 5 different treatments (A, B, C, D, E) according to the sequence determined by randomization. Between each treatment, a minimum of 4 days washout was proposed to minimize any residual nirmatrelvir concentrations prior to start of the next treatment.
  Period 1: Treatment B: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in water under fasted condition.
  Period 2: Treatment A: Single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted condition.
  Period 3: Treatment C: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in infant formula under fasted condition.
  Period 4: Treatment E: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition.
  Period 5: Treatment D: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition.
- Treatment C->B->A->E->D: Each enrolled participant participated in 5 study periods (1-5) to receive 5 different treatments (A, B, C, D, E) according to the sequence determined by randomization. Between each treatment, a minimum of 4 days washout was proposed to minimize any residual nirmatrelvir concentrations prior to start of the next treatment.
  Period 1: Treatment C: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in infant formula under fasted condition.
  Period 2: Treatment B: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in water under fasted condition.
  Period 3: Treatment A: Single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted condition.
  Period 4: Treatment E: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition.
  Period 5: Treatment D: Single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition.
Period: Overall Study
Arm/Group | Treatment A->B->C->D->E | Treatment B->C->A->D->E | Treatment C->A->B->D->E | Treatment A->C->B->E->D | Treatment B->A->C->E->D | Treatment C->B->A->E->D
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in this study.
Groups:
- All Participants: All participants who were enrolled in this study.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 47.2 (8.88)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 4
  45-64 Years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10
  Black or African American | 2

OUTCOME MEASURES:

1. Primary Outcome: AUCinf of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: AUCinf was defined as area under the concentration-time curve from time 0 extrapolated to infinity. AUCinf for nirmatrelvir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve; AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 1, 2, 3, 4, and 5.
Population: All participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted): Participants received a single oral dose of nirmatrelvir 300 (2*150) mg and ritonavir 100 mg tablets under fasted conditions on Day 1 of Periods 1, 2, and 3.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted): Participants received a single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in water under fasted condition on Day 1 of Periods 1, 2, and 3.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted): Participants received a single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in infant formula under fasted condition on Day 1 of Periods 1, 2, and 3.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted): Participants received a single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fasted condition on Day 1 of Periods 4 and 5.
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed): Participants received a single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in vanilla pudding under fed condition on Day 1 of Periods 4 and 5.
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 27090 (18) | 30650 (22) | 33030 (24) | 34000 (22) | 32810 (18)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted); Reference: Nirmatrelvir/ritonavir 300/100 mg tablets (fasted) Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with water (fasted); Test type: Other — The analysis used a mixed effect model with sequence, period and treatment as fixed effects and participant within a sequence as a random effect for comparison: powder mixed with water (fasted) group versus tablets group; Ratio (%) of Adjusted Geometric Mean = 113.13, 90% CI 2-sided [102.77 to 124.53] — The ratios (and 90% confidence Intervals [CIs]) are expressed as percentages
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted); Reference: Nirmatrelvir/ritonavir 300/100 mg tablets (fasted) Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with infant formula (fasted); Test type: Other — The analysis used a mixed effect model with sequence, period and treatment as fixed effects and participant within a sequence as a random effect for comparison: powder mixed with infant formula (fasted) group versus tablets group; Ratio (%) of Adjusted Geometric Mean = 121.91, 90% CI 2-sided [110.75 to 134.20] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted); Reference: Nirmatrelvir/ritonavir 300/100 mg tablets (fasted) Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding (fasted); Test type: Other — The analysis used a mixed effect model with treatment as a fixed effect and participant as a random effect for comparison: powder mixed with vanilla pudding (fasted) group versus tablets group; Ratio (%) of Adjusted Geometric Mean = 125.49, 90% CI 2-sided [114.43 to 137.61] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); Reference: Nirmatrelvir/ritonavir 300/100 mg tablets (fasted) Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding (fed); Test type: Other — The analysis used a mixed effect model with treatment as a fixed effect and participant as a random effect for comparison: powder mixed with vanilla pudding (fed) group versus tablets group; Ratio (%) of Adjusted Geometric Mean = 121.09, 90% CI 2-sided [110.42 to 132.79] — The ratios (and 90% CIs) are expressed as percentages

2. Primary Outcome: AUClast of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for nirmatrelvir was calculated by linear/log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng*hr/mL | 26500 (20) | 30110 (23) | 32470 (25) | 33540 (22) | 32410 (19)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 113.62, 90% CI 2-sided [102.96 to 125.40] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Mean = 122.53, 90% CI 2-sided [111.02 to 135.22] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) of Adjusted Geometric Mean = 126.55, 90% CI 2-sided [115.00 to 139.27] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; Ratio (%) of Adjusted Geometric Mean = 122.28, 90% CI 2-sided [111.11 to 134.57] — The ratios (and 90% CIs) are expressed as percentages

3. Primary Outcome: Cmax of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: Cmax was defined maximum observed concentration. Cmax for nirmatrelvir was observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL | 2862 (20) | 3156 (26) | 4034 (23) | 4287 (22) | 4208 (23)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 110.28, 90% CI 2-sided [99.01 to 122.82] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Mean = 140.97, 90% CI 2-sided [126.57 to 157.01] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) of Adjusted Geometric Mean = 149.83, 90% CI 2-sided [132.86 to 168.96] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; Ratio (%) of Adjusted Geometric Mean = 147.05, 90% CI 2-sided [130.40 to 165.83] — The ratios (and 90% CIs) are expressed as percentages

4. Primary Outcome: AUCinf of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: AUCinf was defined as area under the concentration-time curve from time 0 extrapolated to infinity. AUCinf for ritonavir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve; AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 12
ng*hr/mL | 4005 (37) | 3876 (34) | 3479 (40) | 3986 (34) | 3176 (30)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 96.76, 90% CI 2-sided [87.31 to 107.23] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Mean = 86.86, 90% CI 2-sided [78.38 to 96.26] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) of Adjusted Geometric Mean = 99.29, 90% CI 2-sided [87.39 to 112.80] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; Ratio (%) of Adjusted Geometric Mean = 79.29, 90% CI 2-sided [70.07 to 89.73] — The ratios (and 90% CIs) are expressed as percentages

5. Primary Outcome: AUClast of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for ritonavir was calculated by linear/log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng*hr/mL | 3818 (38) | 3663 (35) | 3303 (40) | 3371 (49) | 2959 (32)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 95.92, 90% CI 2-sided [86.45 to 106.44] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Mean = 86.50, 90% CI 2-sided [77.96 to 95.98] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) of Adjusted Geometric Mean = 88.29, 90% CI 2-sided [72.97 to 106.83] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; Ratio (%) of Adjusted Geometric Mean = 77.49, 90% CI 2-sided [64.04 to 93.76] — The ratios (and 90% CIs) are expressed as percentages

6. Primary Outcome: Cmax of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: Cmax was defined maximum observed concentration. Cmax for ritonavir was observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL | 398.4 (47) | 406.1 (46) | 368.1 (52) | 386.6 (66) | 280.7 (35)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 101.92, 90% CI 2-sided [87.71 to 118.44] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Mean = 92.40, 90% CI 2-sided [79.52 to 107.38] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) of Adjusted Geometric Mean = 97.04, 90% CI 2-sided [78.40 to 120.10] — The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; Ratio (%) of Adjusted Geometric Mean = 70.45, 90% CI 2-sided [56.92 to 87.19] — The ratios (and 90% CIs) are expressed as percentages

7. Secondary Outcome: AUCinf of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir Mixed With Vanilla Pudding Under Fasted/Fed Conditions
Description: AUCinf was defined as area under the concentration-time curve from time 0 extrapolated to infinity. AUCinf for nirmatrelvir (under fasted/fed conditions) was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve; AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 4 and 5.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 34000 (22) | 32810 (18)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); Reference: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding (fasted) Test: Nirmatrelvir/ritonavir 300/100 mg oral powder mixed with vanilla pudding (fed); Test type: Other — The analysis used a mixed effect model with sequence, period and treatment as fixed effects and participant within a sequence as a random effect; Ratio (%) of Adjusted Geometric Mean = 96.50, 90% CI 2-sided [90.08 to 103.37] — The ratios (and 90% CIs) are expressed as percentages

8. Secondary Outcome: AUClast of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir Mixed With Vanilla Pudding Under Fasted/Fed Conditions
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for nirmatrelvir (under fasted/fed conditions) was calculated by linear/log trapezoidal method.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 4 and 5.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 33540 (22) | 32410 (19)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 7, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 96.63, 90% CI 2-sided [90.13 to 103.59] — The ratios (and 90% CIs) are expressed as percentages

9. Secondary Outcome: Cmax of Nirmatrelvir Following the Administration of Nirmatrelvir/Ritonavir Mixed With Vanilla Pudding Under Fasted/Fed Conditions
Description: Cmax was defined maximum observed concentration. Cmax for nirmatrelvir (under fasted/fed conditions) was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 4 and 5.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12
ng/mL | 4287 (22) | 4208 (23)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 7, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 98.15, 90% CI 2-sided [87.28 to 110.36] — The ratios (and 90% CIs) are expressed as percentages

10. Secondary Outcome: AUCinf of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir Mixed With Vanilla Pudding Under Fasted/Fed Conditions
Description: AUCinf was defined as area under the concentration-time curve from time 0 extrapolated to infinity. AUCinf for ritonavir (under fasted/fed conditions) was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve; AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 4 and 5.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 11 | 12
ng*hr/mL | 3986 (34) | 3176 (30)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 7, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 78.49, 90% CI 2-sided [72.42 to 85.07] — The ratios (and 90% CIs) are expressed as percentages

11. Secondary Outcome: AUClast of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir Mixed With Vanilla Pudding Under Fasted/Fed Conditions
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for ritonavir (under fasted/fed conditions) was calculated by linear/log trapezoidal method.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 4 and 5.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 3371 (49) | 2959 (32)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 7, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 87.77, 90% CI 2-sided [69.45 to 110.92] — The ratios (and 90% CIs) are expressed as percentages

12. Secondary Outcome: Cmax of Ritonavir Following the Administration of Nirmatrelvir/Ritonavir Mixed With Vanilla Pudding Under Fasted/Fed Conditions
Description: Cmax was defined maximum observed concentration. Cmax for ritonavir (under fasted/fed conditions) was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after dose on Day 1 of Periods 4 and 5.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12
ng/mL | 386.6 (66) | 280.7 (35)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) vs Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed); [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 7, analysis 1]; Ratio (%) of Adjusted Geometric Mean = 72.60, 90% CI 2-sided [56.87 to 92.68] — The ratios (and 90% CIs) are expressed as percentages

13. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study intervention and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. TEAEs included SAEs and all non-SAEs that occurred during the study.
Time Frame: Baseline up to 28 days after last dose of study intervention (ie, up to 48 days).
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants
  Participants with all-causality TEAEs | 2 | 4 | 5 | 2 | 2
  Participants with all-causality SAEs | 0 | 0 | 0 | 0 | 0
  Participants with treatment-related TEAEs | 2 | 3 | 1 | 1 | 1
  Participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: The following laboratory test abnormalities (without regard to baseline abnormality) were reported during the study: monocytes/leukocytes (percentage [%]) is larger than (>) 1.2x upper limit of normal (ULN), specific gravity (scalar) >1.030, and urine hemoglobin was larger or equal to (>=) 1.
Time Frame: Baseline up to Day 4 of Period 5 (approximately 20 days)
Population: All participants who took at least 1 dose of study intervention and with at least 1 observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants
  Monocytes/Leukocytes (%) >1.2x ULN: number analyzed (Participants) | 12 | 12 | 12 | 6 | 6
  Monocytes/Leukocytes (%) >1.2x ULN | 0 | 0 | 0 | 3 | 2
  Specific gravity (scalar) >1.030: number analyzed (Participants) | 12 | 12 | 12 | 6 | 6
  Specific gravity (scalar) >1.030 | 0 | 0 | 0 | 1 | 0
  Urine hemoglobin >=1: number analyzed (Participants) | 12 | 12 | 12 | 6 | 6
  Urine hemoglobin >=1 | 0 | 0 | 0 | 2 | 1

15. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Supine blood pressure and pulse rate were measured with the participant's arm supported at the level of the heart and recorded after approximately 5 minutes of rest. Vital signs were done predose, 2 hours and 6 hours post dose on Day 1 of each treatment period and also on Day 4 of Period 5. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to Day 4 of Period 5 (approximately 20 days).
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant 12-Lead Electrocardiogram (ECG) Values
Description: A single 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QT, and QTc intervals and QRS complex. All scheduled ECGs were performed after the participant has rested quietly for at least 5 minutes in a supine position. Clinical significance of ECG values was determined at the investigator's discretion.
Time Frame: Baseline up to Day 4 of Period 5 (approximately 20 days).
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination (PE) Values
Description: A complete physical examination included, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A brief physical examination included, at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant reported symptoms.
  Completed PE were performed by trained medical personnel at the investigator site at Screening or Period 1 Day 1 only. A brief PE might be performed at other designated time points at the discretion of the investigator. Clinical significance of physical examination values was determined at the investigator's discretion.
Time Frame: Screening, Baseline up to Day 4 of Period 5 (approximately 20 days).
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Taste Assessment of Mouth Feel After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: The sensory attributes of nirmatrelvir/ritonavir oral powder were evaluated by the participant using a Palatability Questionnaire. Each participant complete the palatability survey immediately following dosing (within 1 min) and at 5, 10, and 20 minutes post oral administration of nirmatrelvir/ritonavir oral powder. For the taste assessment of the study, the data used in the analysis were transcribed and rescaled to a score from 0 (good) to 100 (bad) from the raw measurements on the questionnaire.
Time Frame: 1, 5, 10 and 20 minutes after tasting each study intervention on Day 1 of each period.
Population: All participants who took at least 1 dose of study intervention.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Groups:
- Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted): Participants received a single oral dose of nirmatrelvir 300 mg and ritonavir 100 mg oral powder mixed in water under fasted condition on Day 1 of Periods 1, 2. and 3.
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted)
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  1 minute | 66.8 [54.08 to 79.42] | 65.4 [55.79 to 75.05] | 56.3 [46.17 to 66.50]
  5 minutes | 73.8 [62.36 to 85.14] | 60.3 [51.86 to 68.64] | 57.2 [48.16 to 66.17]
  10 minutes | 72.4 [61.34 to 83.49] | 59.3 [52.22 to 66.28] | 56.7 [46.44 to 66.89]
  20 minutes | 65.5 [55.87 to 75.13] | 56.3 [46.43 to 66.24] | 53.4 [43.30 to 63.54]

19. Secondary Outcome: Taste Assessment of Bitterness After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 18
Time Frame: 1, 5, 10 and 20 minutes after tasting each study intervention on Day 1 of each period.
Population: All participants who took at least 1 dose of study intervention.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted)
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  1 minute | 75.3 [62.27 to 88.23] | 72.0 [63.22 to 80.78] | 61.4 [51.35 to 71.49]
  5 minutes | 75.4 [65.00 to 85.83] | 66.5 [59.09 to 73.91] | 58.2 [50.21 to 66.12]
  10 minutes | 72.1 [62.72 to 81.44] | 56.8 [47.15 to 66.35] | 56.8 [46.59 to 67.08]
  20 minutes | 66.2 [56.47 to 75.86] | 57.0 [48.14 to 65.86] | 55.4 [43.97 to 66.86]

20. Secondary Outcome: Taste Assessment of Tongue/Mouth Burn After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 18
Time Frame: 1, 5, 10 and 20 minutes after tasting each study intervention on Day 1 of each period.
Population: All participants who took at least 1 dose of study intervention.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted)
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  1 minute | 31.3 [17.50 to 45.00] | 36.3 [20.15 to 52.52] | 32.4 [16.58 to 48.25]
  5 minutes | 33.9 [18.74 to 49.09] | 29.9 [16.51 to 43.32] | 29.8 [14.73 to 44.93]
  10 minutes | 36.3 [19.61 to 52.89] | 29.7 [17.17 to 42.17] | 29.7 [15.83 to 43.50]
  20 minutes | 31.0 [17.22 to 44.78] | 25.8 [12.18 to 39.49] | 26.7 [13.46 to 39.87]

21. Secondary Outcome: Taste Assessment of Throat Burn After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 18
Time Frame: 1, 5, 10 and 20 minutes after tasting each study intervention on Day 1 of each period.
Population: All participants who took at least 1 dose of study intervention.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted)
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  1 minute | 30.9 [17.52 to 44.31] | 31.7 [15.42 to 47.92] | 26.4 [12.35 to 40.48]
  5 minutes | 34.5 [18.32 to 50.68] | 37.5 [21.44 to 53.56] | 27.3 [12.56 to 41.94]
  10 minutes | 34.4 [18.62 to 50.21] | 34.8 [17.90 to 51.60] | 29.4 [15.89 to 42.95]
  20 minutes | 33.7 [18.90 to 48.43] | 31.3 [16.10 to 46.40] | 27.8 [13.96 to 41.54]

22. Secondary Outcome: Taste Assessment of Overall Liking After Administration of Nirmatrelvir/Ritonavir in Different Delivery Vehicles
Description: as for outcome 18
Time Frame: 1, 5, 10 and 20 minutes after tasting each study intervention on Day 1 of each period.
Population: All participants who took at least 1 dose of study intervention.
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted)
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale
  1 minute | 73.5 [62.24 to 84.76] | 65.0 [53.60 to 76.40] | 55.8 [45.43 to 66.24]
  5 minutes | 74.7 [64.19 to 85.15] | 66.3 [54.81 to 77.69] | 55.9 [46.29 to 65.54]
  10 minutes | 72.6 [63.09 to 82.08] | 62.4 [53.45 to 71.39] | 57.1 [47.06 to 67.11]
  20 minutes | 64.7 [51.68 to 77.66] | 56.4 [42.48 to 70.35] | 56.3 [46.25 to 66.42]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study intervention (ie, up to 48 days).
Arm/Group | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 4/12 | 5/12 | 2/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir/Ritonavir 300/100 mg Tablets (Fasted) (N=12) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Water (Fasted) (N=12) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Infant Formula (Fasted) (N=12) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fasted) (N=12) | Nirmatrelvir/Ritonavir 300/100 mg Oral Powder Mixed With Vanilla Pudding (Fed) (N=12)
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 1 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT05544786/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT05544786/SAP_001.pdf